CLINICAL TRIAL: NCT05334680
Title: Wearable Sensor to Monitor and Track COVID-19-like Signs and Symptoms to Develop Better Care Strategies for COVID-19 Pandemic - An Exploratory Study
Brief Title: International Validation of Wearable Sensor to Monitor COVID-19 Like Signs and Symptoms
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Arun Jayaraman, PT, PhD (Other)
Collaborators: United States - India Science and Technology Endowment Fund (Unknown); Northwestern University (Other); Induss Hospitals (Unknown); Bionic Yantra (Unknown); Clinfinite Solutions (Network); Indian Institute of Technology Kharagpur (Unknown)
Responsible Party: Sponsor-Investigator, Arun Jayaraman, PT, PhD, Director Max Nader Laboratory, Shirley Ryan AbilityLab
Organization: Shirley Ryan AbilityLab (Other)
Other Study IDs: BY/001/2021
Record Dates: First submitted 2022-04-15; First posted 2022-04-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: Wearable sensor; Machine learning; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Individuals experiencing COVID-19 like symptoms.
  Interventions: Device: ANNE Sensor
- Healthy Controls: Individuals without any known significant health problems
  Interventions: Device: ANNE Sensor

INTERVENTIONS:
Device: ANNE Sensor — The data collected from this sensor contains a wide range of core and novel respiratory digital biomarkers as a home-based early identification system. The core measurements include: heart rate, heart rate variability, temperature, physical activity (including sleep quality) and respiratory rate. The novel respiratory digital biomarkers include: respiratory cadence (expiration / inspiration time), coughing, swallowing, throat clearing, and talk time.

SUMMARY:
1. Deploy wearable COVID sensor to collect high resolution physiological data (temperature, cardiac, respiratory and physical activity) from COVID positive patients.
2. Use collected data to train algorithm for assessing the risk of individuals presenting with symptoms suggestive of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-95 years old
* Currently experiencing any COVID-like signs and symptoms such as fever, cough, shortness of breath, trouble breathing, persistent pain or pressure in the chest, confusion or inability to arouse, bluish lips or face.
* Individuals who are not experiencing any COVID like signs and symptoms (will be asked to be healthy control)
* Able and willing to give written consent and comply with study procedures.

Exclusion Criteria:

* Inability to understand instructions and follow a three step command.
* The subject is pregnant, nursing or planning a pregnancy.
* Inability to provide written consent.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who may have experienced COVID-19 like symptoms.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-03-08 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | Baseline; Possible reassessment up to five days after consent
  Instantaneous heart rate associated with various activity levels
Respiratory frequency | Baseline; Possible reassessment up to five days after consent
  Participants will be asked to breathe normally before and after walking for 30 seconds.
Cough Frequency | Baseline; Possible reassessment up to five days after consent
  Cough signal characteristics during five consecutive coughs
Body temperature | Baseline; Possible reassessment up to five days after consent
  Periodic temperature readings throughout the activity sequence

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (3):
- India (3):
  - St. Georges Hospital, Mumbai, Maharashtra
  - Lifepoint Multi-Specialty Hospital, Pune, Maharashtra
  - Induss Hospitals, Hyderabad, Telangana